CLINICAL TRIAL: NCT02233335
Title: The Factors Associated With the Recurrence in Patients With Cushing Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201305026RINC
Record Dates: First submitted 2014-08-27; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Cushing Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cushing syndrome refers the manifestations induced by chronic glucocorticoid excess and may arise from various causes. Iatrogenic Cushing syndrome accounts for most patients, when they are given exogenous glucocorticoid treatment. In contrast, spontaneous Cushing syndrome results from endogenous glucocorticoid over-secretion. Although Cushing disease is rare, it is the most common cause of spontaneous Cushing syndrome. The patient with Cushing disease has a pituitary corticotroph adenoma, which overproduces adrenocorticotropic hormone (ACTH). ACTH then stimulates adrenal gland to over-secret glucocorticoid. Patients with untreated Cushing disease were shown to have poor prognosis, estimated a 5-year survival rate of 50%. The first line treatment is tumor resection. Other managements include radiotherapy, medication and bilateral adrenalectomy. The initial remission rate is high (66-90%). However, some patients encounter with disease recurrence during follow-up.

The aim of this study is to clarify the factors associated with the recurrence after treatment. In this study, we will review the patients with Cushing disease thoroughly and analyze associated predisposing factors. These risk factors can remind the clinical physician to early detect the recurrent disease in these patients, and further prevent morbidity and mortality in their later lives.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed Cushing's disease

Exclusion Criteria:

* Already received treatment in other hospital
* Ectopic Cushing's syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cushing's disease who presented to the National Taiwan University Hospital between 1992 and 2011
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with disease persistence or recurrence after surgery, which was determined by clinical symptoms, biochemical lab, dynamic test and image study | participants were followed at 3 months after treatment for short-term outcome measure and followed until the last hospital visit, an average of 4.7 years, for long-term outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Chun Chang, M.D., Ph.D., Study Chair — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] PLOTZ CM, KNOWLTON AI, RAGAN C. The natural history of Cushing's syndrome. Am J Med. 1952 Nov;13(5):597-614. doi: 10.1016/0002-9343(52)90027-2. No abstract available. PMID 12996538
- [Background] Etxabe J, Vazquez JA. Morbidity and mortality in Cushing's disease: an epidemiological approach. Clin Endocrinol (Oxf). 1994 Apr;40(4):479-84. doi: 10.1111/j.1365-2265.1994.tb02486.x. PMID 8187313
- [Background] Swearingen B, Biller BM, Barker FG 2nd, Katznelson L, Grinspoon S, Klibanski A, Zervas NT. Long-term mortality after transsphenoidal surgery for Cushing disease. Ann Intern Med. 1999 May 18;130(10):821-4. doi: 10.7326/0003-4819-130-10-199905180-00015. PMID 10366371
- [Background] Lindholm J, Juul S, Jorgensen JO, Astrup J, Bjerre P, Feldt-Rasmussen U, Hagen C, Jorgensen J, Kosteljanetz M, Kristensen L, Laurberg P, Schmidt K, Weeke J. Incidence and late prognosis of cushing's syndrome: a population-based study. J Clin Endocrinol Metab. 2001 Jan;86(1):117-23. doi: 10.1210/jcem.86.1.7093. PMID 11231987
- [Background] Hammer GD, Tyrrell JB, Lamborn KR, Applebury CB, Hannegan ET, Bell S, Rahl R, Lu A, Wilson CB. Transsphenoidal microsurgery for Cushing's disease: initial outcome and long-term results. J Clin Endocrinol Metab. 2004 Dec;89(12):6348-57. doi: 10.1210/jc.2003-032180. PMID 15579802
- [Background] Dekkers OM, Biermasz NR, Pereira AM, Roelfsema F, van Aken MO, Voormolen JH, Romijn JA. Mortality in patients treated for Cushing's disease is increased, compared with patients treated for nonfunctioning pituitary macroadenoma. J Clin Endocrinol Metab. 2007 Mar;92(3):976-81. doi: 10.1210/jc.2006-2112. Epub 2007 Jan 2. PMID 17200171
- [Background] Clayton RN, Raskauskiene D, Reulen RC, Jones PW. Mortality and morbidity in Cushing's disease over 50 years in Stoke-on-Trent, UK: audit and meta-analysis of literature. J Clin Endocrinol Metab. 2011 Mar;96(3):632-42. doi: 10.1210/jc.2010-1942. Epub 2010 Dec 30. PMID 21193542
- [Background] Hassan-Smith ZK, Sherlock M, Reulen RC, Arlt W, Ayuk J, Toogood AA, Cooper MS, Johnson AP, Stewart PM. Outcome of Cushing's disease following transsphenoidal surgery in a single center over 20 years. J Clin Endocrinol Metab. 2012 Apr;97(4):1194-201. doi: 10.1210/jc.2011-2957. Epub 2012 Jan 25. PMID 22278423
- [Background] Atkinson AB, Kennedy A, Wiggam MI, McCance DR, Sheridan B. Long-term remission rates after pituitary surgery for Cushing's disease: the need for long-term surveillance. Clin Endocrinol (Oxf). 2005 Nov;63(5):549-59. doi: 10.1111/j.1365-2265.2005.02380.x. PMID 16268808
- [Background] Pikkarainen L, Sane T, Reunanen A. The survival and well-being of patients treated for Cushing's syndrome. J Intern Med. 1999 May;245(5):463-8. doi: 10.1046/j.1365-2796.1999.00483.x. PMID 10363746